CLINICAL TRIAL: NCT05749692
Title: The Impact of COVID-19 Infection on the Symptoms of Functional Dyspepsia
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Air Force Military Medical University, China (Other)
Responsible Party: Principal Investigator, Yanglin Pan, professor, Air Force Military Medical University, China
Other Study IDs: KY20221243-F-1
Record Dates: First submitted 2023-02-28; First posted 2023-03-01 (Actual); Last update posted 2023-03-01 (Actual); Status verified 2023-02

CONDITIONS: Dyspepsia
Keywords: Functional Dyspepsia; COVID-19
MeSH Terms: conditions — Dyspepsia; COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- The COVID-19 infected group: Functional dyspepsia patients infected with COVID-19

SUMMARY:
Although respiratory symptoms were predominant in patients infected with COVID-19, gastrointestinal symptoms were always reported in about 10% patients. Previous studies demonstrated that the SARS-CoV-2 virus still persists in stool samples for a long time after initial infection. Moreover, some patients had a longer duration of COVID-19-related gastrointestinal symptoms, which was defined as "post-acute COVID-19 syndrome".

Previous studies have shown that functional gastrointestinal disorders may occur after acute gastroenteritis. Functional dyspepsia (FD) is one of the most common functional gastrointestinal disorders. FD was reported to be correlated with multiple pathophysiological mechanisms, including GI bacterial imbalance, disordered gut microbiota, and disturbed barrier and immune function. It is unknown whether COVID-19 infection could exacerbate the symptoms of FD. Therefore, we followed up a group of FD patients before and after COVID-19 and investigate the impact of COVID-19 infection on the symptoms of FD.

ELIGIBILITY:
Inclusion Criteria:

1. aged ≥18 years old
2. Patients who met broad criteria of dyspepsia before infection

Exclusion Criteria:

1. organ failure defined by Marshall standard
2. severe psychiatric illnesses
3. suspected or identified bowel obstruction
4. known malignancy
5. pregnancy or lactation
6. unable to provide consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients aged ≥ 18 years old who met broad criteria of dyspepsia were eligible for our study before infection.
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2022-12-01 (Actual); Primary Completion 2023-08-01 (Estimated); Study Completion 2023-08-01 (Estimated)

PRIMARY OUTCOMES:
a score of 1 or 2 (extremely worse) on a 7-Likert scale assessing dyspepsia symptom change | 1month, 3 months, 6 months
  The patients were interviewed to answer the question "Compared with condition before infection, how about is your gut condition now?" The following questions were chosen: (1) extremely worse, (2) worse, (3) slightly worse, (4) same as before, (5) slightly better, (6) better or (7) much better.

SECONDARY OUTCOMES:
Global Overall Symptom score (GOSS) | 1month, 3 months, 6 months
  The GOSS consists of 10 cardinal items (epigastric pain, epigastric discomfort, Heartburn, acid regurgitation, upper abdominal bloating, belching, nausea, early satiety, postprandial fullness, other epigastric symptoms(eg. epigastric burning). Each item can be scored from 1 (no) to 7 (worst).
subtypes of functional dyspepsia | 6 months
  functional dyspepsia was classified into three subgroups：(1) Postprandial Distress Syndrome, defined as Bothersome postprandial fullness or/and Bothersome early satiation. (2) Bothersome epigastric pain AND/OR Bothersome epigastric burning. (3) mixed syndrome, defined when postprandial distress syndrome and epigastric pain syndrome presented simultaneously.
self-reported severity of symptoms by patients | 1month, 3 months, 6 months
  patients rated the severity of FD as mild, moderate, and severe
Other gastrointestinal symptoms | 1month, 3 months, 6 months
  Recurrent lower abdominal pain， dysphoria， altered bowel habit， stool character change， etc.
Short Form of Nepean Dyspepsia Index (SF-NDI) | 1month, 3 months, 6 months
  The SF-NDI consists of 10 questions regarding the effects of dyspepsia symptoms ("stomach problems") on different aspects of life (tension, interference with daily activities, eating/drinking, knowledge/control, and work/study). Each response can be from 1 (not at all affected) to 5 (extremely affected), or 0 (N/A), for a total summed score out of 50.
Hospital anxiety and depression scale | 1month, 3 months, 6 months
  Anxiety and depression of patients are assessed by using Hospital Anxiety and Depression Scale.It contains 14 items (7 anxiety and 7 depression), which assess symptoms experienced during the past week on a 0-3 scale. A subscore of > 8 for depression or anxiety would indicate a clinical case.

CONTACTS AND LOCATIONS:
Locations (1):
- Xijing Hospital of Digestive Diseases, Xi'an, Shaanxi, China